CLINICAL TRIAL: NCT03023774
Title: Effects of Granulocyte Colony-stimulating Factor (GCSF)-Neupogen on Cases With Thin Endometrium or Previous Implantation Failure in ICSI Cycles
Brief Title: Use of Gcsf in Patients With Recurrent Ivf/Icsi Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Dr wessam magdi abuelghar, principal investigator, Ain Shams Maternity Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ABT-1233-RV
Record Dates: First submitted 2017-01-12; First posted 2017-01-18 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Fertility Disorders
MeSH Terms: interventions — Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- neupogen (Other): neupogen (granulocyte colony-stimulating factor) 30 IU once intrauterine at the time of ovum pickup
  Interventions: Drug: Neupogen

INTERVENTIONS:
Drug: Neupogen — neupogen 30 IU once intrauterine at the time of ovum pickup
  Other Names: granulocyte colony-stimulating factor

SUMMARY:
Evaluate the effectiveness of granulocyte colony-stimulating factor (GCSF) in the treatment of thin endometrium or in women with recurrent implantation failure in ICSI cycles

DETAILED DESCRIPTION:
Prospective analytical study which will be conducted at a private IVF center starting from june 2016.

the study will be recruited from both the fertility clinics and centers by fulfilling inclusion and exclusion criteria , all patient will be subjected to complete history taking medical and fertility history including previous induction or implantation failure.

patients will be randomized into two groups, group A will be treated with neupogen 30 international unit (IU) and group B will be treated with clexane 40mg and estrogen.

study procedure: ovaries were stimulated with standard protocol (long GnRH Agonist) or gonadotrophic releasing hormone (GnRH Antagonist, when at least 3 follicles achieved 18 mm diameter, Human chorionic gonadotrophic (hCG) (10000 IU) was administered for ovulation triggering, transvaginal oocyte retrieval was performed at 36-38 hours after injection of hCG . the oocytes were fertilized by intracytoplasmic sperm injection (ICSI) method. the thickness of endometrium was evaluated on the day of oocyte retrieval and syringe which containing (300 mcg/1 ml) GCSF (neupogen) was infused slowly in the uterine cavity and after 5 days (before embryo transfer) endometrial thickness was evaluated again. all patients received oral and parenteral progesterone for luteal phase support.

ELIGIBILITY:
Inclusion Criteria:

* male partner with normal semen analysis according to world health organization (WHO) 2010.
* female partner under the age of 36 presented with: a-thin endometrium (less 7 mm on transvaginal ultrasound) or b- previous history multiple unexplained
* female with no history of Asherman's syndrome , fibroids, and polyps in diagnostic hysteroscopy

Exclusion Criteria:

* women with sickle cell disease, renal insufficiency, upper respiratory infection or pneumonia, chronic neutropenia, known past or present malignancy

Max Age: 36 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Actual)
Dates: Start 2016-06; Primary Completion 2016-10 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
increase in endometrial thickness (above 7 mm) | one week

SECONDARY OUTCOMES:
chemical pregnancy (serum beta hCG titre more than (25 mili liter international unit (mIU)/ml) and clinical pregnancy defined as the presence of an intrauterine gestational sac on transvaginal ultrasound (TVS)as 6 weeks. | 6 week

IPD SHARING:
Plan to Share IPD: Yes
Female 35 years maximum have failed icsi due to low endometrium thickness